ACE-WIVI-001

Statistical Analysis Plan

Version 2.0, dated: 31 January 2018

Protocol Number: ACE-WM-001

Protocol Title: An Open-label, Phase 2 Study of ACP196 in Subjects with

Waldenström Macroglobulinemia

Version: 2.0

Version date: 31 January 2018

The undersigned have reviewed this plan and find it to be consistent with the requirements of the protocol as it applies to their respective areas



#### CONFIDENTIAL

This document (and all copies thereof) is the property of Acerta Pharma and contains valuable trade secrets and confidential information, including proprietary technical and business information. By accepting this document, you agree that the Confidential Information contained herein will not be disclosed to others without prior written authorization from Acerta Pharma and shall only be used for the purposes intended by the document.

# **Statistical Analysis Plan**

An Open-label, Phase 2 Study of ACP-196 in Subjects with Waldenström Macroglobulinemia

**Protocol Number: ACE-WM-001** 

Version: Date:

**Study Statistician:** 



Acerta Pharma 

# **TABLE OF CONTENTS**

| Table | e of Contents | 2 |
|---|---|---|
| Table | e of Abbreviations | 4 |
| 1. | INTRODUCTION | 6 |
| 2. | OBJECTIVES | 6<br>7 |
| 3. | STUDY OVERVIEW | 7 |
| 4. | STUDY ENDPOINTS | 10<br>10 |
| 5. | ANALYSIS POPULATION | 11 |
| 6. | SUBGROUP ANALYSIS | 11 |
| 7. | INTERIM ANALYSIS | 11 |
| 8. | PRIMARY AND FINAL ANALYSIS AND CLINICAL STUDY REPORT | 12 |
| 9. | MISSING VALUES | 12 |
| 10. | STATISTICAL METHODS OF ANALYSIS 10.1 General Principles 10.2 Subject Accountability 10.3 Important Protocol Deviations 10.4 Baseline Data 10.4.1 Demographics 10.4.2 Baseline Characteristics 10.4.3 Baseline Disease Characteristics 10.5 Treatment and Medications 10.5.1 Prior Anticancer Therapies 10.5.2 Concomitant Medications 10.5.3 Exposure to Study Drug 10.6 Analyses of Efficacy Endpoints | 13<br>13<br>14<br>14<br>15<br>15 |
| | 10.6.1 Definition of Primary Endpoints | |

| | 10.6.3 | Definition of Secondary Endpoints | 16 |
|---|---|---|---|
| | 10.6.4 | Analysis Method for Secondary Endpoints | 17 |
| | 10.7 Analyse | es Safety Endpoints | 19 |
| | 10.7.1 | Adverse Events | 19 |
| | 10.7.2 | Adverse Events of Clinical Interest | 19 |
| | 10.7.3 | Laboratory Test Results | 20 |
| | 10.7.4 | Vital Signs | 20 |
| | 10.7.5 | Eastern Cooperative Oncology Group (ECOG) Performance Status | 20 |
| | 10.7.6 | Electrocardiogram (ECG) | 20 |
| 11. | CHANGES F | ROM PROTOCOL-SPECIFIED ANALYSES | 20 |
| 12. | LITERATUR | E CITATIONS / REFERENCES | 21 |
| 13. | APPENDICE | S | 22 |
| | 13.1 Definition | ons | 22 |
| | 13.1.1 | Study Day | 22 |
| | 13.1.2 | Baseline Value and Post-baseline Value | 22 |
| | 13.1.3 | Duration of Treatment and Time on Study | 22 |
| | 13.1.4 | Average Daily Dose and Relative Dose Intensity | 22 |
| | 13.1.5 | Age | 23 |
| | 13.1.6 | Year and Month | 23 |
| | 13.1.7 | Treatment-emergent Adverse Events | 23 |
| | 13.1.8 | Refractory Disease | 23 |
| | 13.1.9 | Extrameduallary Disease, Bone Marrow Involvement and Advanced Disease at Baseline | 23 |
| | 13.2 Imputat | tion Rules for Partial or Missing Dates | 23 |
| | | ing Rules | |
| | | s Windows for EORTC QLQ-30 | |

ACE-WM-001

**Statistical Analysis Plan** 

Version 2.0, dated: 31 January 2018

### **TABLE OF ABBREVIATIONS**

ACP-196 acalabrutinib

AE(s) adverse event(s)

AMA American medical association

ANC absolute neutrophil count

BID twice per day

CI confidence interval

CR complete response (remission)

CRF case report form

CSR clinical study report

CTCAE common terminology criteria for adverse events

DOR duration of response ECG electrocardiogram

ECOG eastern cooperative oncology group

EORTC european organization for research and treatment of cancer

HGB hemoglobin

IRC independent review committee
IPD important protocol deviation

MCL mantle cell lymphoma

MedDRA medical dictionary for regulatory activities

MR minor response

NCI national cancer institute
NDA new drug application
ORR overall response rate

OS overall survival

PD progressive disease PD pharmacodynamics

PFS progression-free survival

PK pharmacokinetics

PLT platelet

PR partial response

PRO patient reported outcome

PT preferred term
QD once per day

QLQ-C30 core quality of life questionnaire

Acerta Pharma 

ACE-WM-001 Statistical Analysis Plan

Version 2.0, dated: 31 January 2018

QTc corrected QT interval R/R relapsed/refractory

SAE(s) serious adverse event(s) SAP statistical analysis plan

SD stable disease

SI the international system of units

SOC system organ class

TEAE(s) treatment-emergent adverse events

VGPR very good partial response
WHO world health organization

WM waldenström macroglobulinemia

Acerta Pharma 

# 1. INTRODUCTION

| This statistical analysis plan (SAP) provides details of efficacy and safety analyses that |
|---|
| have been outlined within ACE-WM-001 , which is entitled "An |
| Open-label, Phase 2 Study of ACP-196 in Subjects with Waldenström |
| Macroglobulinemia" |

Hereafter, acalabrutinib (a generic name for ACP-196) will be used in place of ACP-196 in this document.

Separate reports will be generated for pharmacokinetic (PK) and pharmacodynamics (PD) data.

The analysis will be executed by the biometrics department of Acerta Pharma unless otherwise specified.

#### 2. OBJECTIVES

# 2.1 Primary Objectives

The primary objective of this study is to:

 To determine the ORR of acalabrutinib in subjects with WM as assessed by investigator.

Acerta Pharma 

# 2.2 Secondary Objectives

The secondary objectives are as follows:

- To determine the ORR of acalabrutinib by IRC
- To determine the DOR of acalabrutinib by investigator and by IRC, respectively
- To determine the PFS of acalabrutinib by investigator and by IRC, respectively
- To determine the overall survival (OS) of acalabrutinib
- To characterize the PK profile of acalabrutinib
- To characterize the safety of acalabrutinib
- To evaluate the effect of acalabrutinib in health-related quality of life

# 2.3 Exploratory Objective

To evaluate the PD effects of acalabrutinib

#### 3. STUDY OVERVIEW

# 3.1 Study Design

This study is a multicenter open-label clinical trial evaluating the safety and efficacy of acalabrutinib 100 mg twice a day (BID) in subjects with previously treated WM using a Simon's optimal two-stage design. In addition, a small cohort of subjects with previously untreated WM will be enrolled as an exploratory cohort to determine the preliminary safety and efficacy of acalabrutinib in this patient population.

Treatment with acalabrutinib may be continued until disease progression (PD) or an unacceptable drug-related toxicity occurs. All subjects who discontinue acalabrutinib will have a safety follow-up visit 30 (+ 7) days after the last dose of study drug to monitor for resolution or progression of adverse event(s) (AEs) and to document the occurrence of any new events, regardless of whether the subject receives a new anticancer therapy or demonstrates PD within this timeframe.

All subjects will have hematology, chemistry, and urinalysis safety panels done at screening. Once dosing commences (Day 1), all subjects will be evaluated for safety, including serum chemistry and hematology, once weekly for the first 4 weeks, every 2 weeks in Cycle 2, monthly thereafter until Cycle 12, and every 3 months after Cycle 12.

Acerta Pharma 

3.2

Sample Size

Version 2.0, dated: 31 January 2018

PK testing will be done in Cycle 1 only, and PD testing will be done in Cycle 1 and Cycle 2. PK/PD will be done on all subjects in the previously untreated cohort and on up to 12 subjects in the previously treated cohort.

Assessments for efficacy will be done at the end of every cycle. For subjects with baseline (screening) extramedullary disease, follow-up radiologic assessments are required at the end of Cycle 2 ( $\pm$  7 days), Cycle 4 ( $\pm$  7 days), Cycle 6 ( $\pm$  7 days), and then every 3 cycles (12 weeks,  $\pm$  7 days) thereafter or more frequently at the investigator's discretion.

A single, independent interim analysis of ORR will be performed when subjects from Stage 1 (28 subjects) are evaluable for response.

The primary analysis defined as all subjects have completed Cycle 27 or have discontinued before Cycle 27.

This study will use an IRC to confirm ORR, DOR and PFS for the final analysis. IRC assessments will not be available for primary analysis.

Acerta Pharma 



In total, 106 subjects were enrolled over a 15-month period. The treatment cohorts are as follows:

| Cohort | Population | Dose | Patient | Enrollment |
|--------|----------------------|------------|----------|------------|
| | | Regimen | Enrolled | Status |
| 1 | Previously treated | 100 mg BID | 86 | Closed |
| | Previously treated | 200 mg QD | 5 | Closed |
| 2 | Previously untreated | 100 mg BID | 14 | Closed |
| | Previously untreated | 200 mg QD | 1 | Closed |

During development of WM-001, this study was designed to test the null hypothesis that the ORR is  $\leq$  35% against the alternative hypothesis that it is  $\geq$  55%. For previously treated WM patients, using Simon's optimal two-stage design, a total sample size of 76 subjects has 90% power to achieve a one-sided significance level of 0.025. In Stage 1, 28 subjects will be evaluated for efficacy. If  $\geq$  12 out of 28 subjects (43%) achieve a response, then the study will continue to full enrollment. In Stage 2, a further 48 subjects will be enrolled. With original Simon's optimal two-stage design, an ORR of  $\geq$  46% (i.e.,  $\geq$  35 subjects responding out of 76 subjects evaluated) will achieve a one-sided significance level of  $\leq$  0.025.

### 4. STUDY ENDPOINTS

# 4.1 Co-primary Endpoints

The co-primary endpoints are:

- ORR, defined as a subject achieving a minor response (MR) or better according to the response assessment criteria for WM (Owen 2013), as assessed by investigators
- ORR, defined as a subject achieving a MR or better according to the response assessment criteria defined by modified 3<sup>rd</sup> IWWM workshop criteria (Kimby 2006), as assessed by investigators

# 4.2 Secondary Endpoints

# Efficacy:

- ORR, defined by modified 3<sup>rd</sup> IWWM workshop criteria (Kimby 2006), as assessed by IRC
- DOR by investigator, assessed using response assessment criteria for WM (Owen 2013) and modified 3<sup>rd</sup> IWWM workshop criteria (Kimby 2006)
- DOR by IRC, assessed using the modified 3<sup>rd</sup> IWWM workshop criteria (Kimby 2006)
- PFS by investigator, assessed using Response Assessment Criteria for WM (Owen 2013) and modified 3<sup>rd</sup> IWWM workshop criteria (Kimby 2006)
- PFS by IRC, assessed using the modified 3<sup>rd</sup> IWWM workshop criteria
- Overall survival (OS)
- Effect of acalabrutinib on peripheral T/B/natural killer (NK) cell counts
- Effect of acalabrutinib on serum immunoglobulin levels

# Safety:

- Frequency, severity, and relatedness of AEs
- Frequency of AEs requiring discontinuation of study drug or dose reductions

#### Pharmacokinetics:

Plasma pharmacokinetics of acalabrutinib

Acerta Pharma 

Patient reported outcomes (PRO):

· Health-related quality of life

# 4.3 Exploratory Endpoints

Pharmacodynamics: BTK occupancy and biologic markers of B-cell function.

# 5. ANALYSIS POPULATION

The analysis population is defined as follows:

**All-treated population**: All enrolled subjects who receive ≥ 1 dose of study drug. The demographics, baseline and disease characteristics, safety analyses and efficacy analyses will be performed on the all-treated population.

All enrolled subjects were treated with at least one dose of study drug in this study, thus all-treated population is the same as the enrolled population.

**Efficacy-evaluable population**: All subjects in the all-treated population who have ≥ 1 evaluable response assessment after the first dose of study drug. Co-primary endpoints and ORR based on IRC assessments will also be performed using efficacy-evaluable population.

#### 6. SUBGROUP ANALYSIS

Subgroup analysis for primary efficacy endpoints and ORR based on IRC assessment using both criteria will be planned for demographics and baseline characteristics as follows:

- Age (< 65 years versus ≥ 65 years)</li>
- ECOG performance status at baseline (0 versus >= 1)
- Number of prior systemic therapies (1 ~ 3 versus > 3)
- Hemoglobin (HGB <= 110 g/L versus HGB > 110 g/L)
- Serum IgM (< 4000 mg/dl versus >= 4000 mg/dl)
- Bone marrow disease involvement (positive/negative/indeterminant)

Subgroup analysis for MYD88 and CXCR4 data will be planned as needed.

# 7. INTERIM ANALYSIS

Acerta Pharma 

An interim analysis for futility based on response rate was performed in September 2015 per protocol amendment 3.0 dated 13March2015. As of the data cut-off on 31August2015, 14 responders were observed among 27 subjects. The required response rate for continuation (≥ 12/28 responders) was exceeded and enrollment continued based on this result.

A safety interim analysis was performed based on data cut-off on 02January2017. An interim safety CSR based on this data was submitted to FDA to support the sponsor's new drug application (NDA) for the treatment of adult patients with mantle cell lymphoma (MCL) who have received at least one prior therapy.

#### 8. PRIMARY AND FINAL ANALYSIS AND CLINICAL STUDY REPORT

The primary analysis will occur when all subjects have completed Cycle 27 or have discontinued before Cycle 27 as per protocol amendment 7.0. A final analysis will be performed at end of study. End of study is defined as 48 cycles after enrollment of last subjects.

Onset of response is expected to be around 2 months. The primary analysis time point corresponds to a minimum of more than 2 years of follow-up for all subjects and it allows time to demonstrate durability of response. Base on the literature, PFS is expected to mature around 4 years and the final analysis time point allows a robust estimate of overall PFS.

#### 9. MISSING VALUES

Safety Data

No imputation of values for missing data will be performed except for missing or partial dates according to prespecified, conservative imputation rules. The algorithm for handling missing or partial dates is provided in Appendix 13.2.

Efficacy Data

Acerta Pharma 

The method for handling missing data is described in the definition for each of the efficacy endpoints. Every effort will be made to obtain complete dates for deaths. In the event of a partial or missing death date, the algorithm in Appendix 13.2 will be used.

#### 10. STATISTICAL METHODS OF ANALYSIS

#### 10.1 **General Principles**

Descriptive statistics will be used to summarize disposition, demographic, baseline characteristics, disease characteristics, prior anticancer therapy, concomitant medication, study drug administration, efficacy and safety outcomes. Descriptive summary of discrete data will present the sample size and the incidence as frequency and percentage. Descriptive summaries of continuous data will present the sample size, group mean, standard deviation, median, and range.

Confidence intervals (CIs), when presented, will generally be constructed at the 95% level. For binomial variables, the exact method for CIs will be employed unless otherwise specified.

Calculation of time to event or duration of event (e.g., DOR) will be based on actual study day of the event rather than nominal visit date.

#### 10.2 Subject Accountability

The number of subjects enrolled by site, country and region (US and ex-US) will be presented. Subject disposition will be summarized for all enrolled subjects including the following information:

- Subject status on study drug
- Count and reason for study drug discontinuation
- Subject status for the study
- Count and reason for study termination
- Time on study

#### 10.3 **Important Protocol Deviations**

The important protocol deviations (IPDs) categories are defined and managed by the study team during the IPD reviews throughout the study before database lock. These

Acerta Pharma 

definitions of IPD categories, sub-category codes and descriptions will be used during the study. The final IPD list is used to produce the summary of IPDs table and the list of subjects with IPDs.

#### 10.4 Baseline Data

### 10.4.1 Demographics

- Age (continuous)
- Age category (< 65 years versus ≥ 65 years)</li>
- Sex (Male, Female)
- Ethnicity
- Race
- Region

#### 10.4.2 Baseline Characteristics

- Height (cm)
- Weight (kg)
- ECOG performance status

### 10.4.3 Baseline Disease Characteristics

- Number of prior systemic therapies (continuous and grouped as 1 ~ 3 versus > 3)
- Time (years) from initial diagnosis to first acalabrutinib dose
- Serum IgM (mg/dl) (continuous and grouped as > 4000 mg/dl))
- Extramedullary disease (yes/no)
- Advanced disease (extrameduallary disease and/or bone marrow involvement) (yes/no)
- Bone marrow involvement (positive/negative/indeterminant)
- Refractory disease at baseline (yes/no)
- Hematology: hemoglobin (HGB), absolute neutrophil counts (ANC), platelet counts (PLT) and absolute lymphocyte counts.

Acerta Pharma 

Clinically meaningful cytopenia (ANC <= 1.5 x 10<sup>9</sup>/L; HGB<=100 g/L; HGB <= 110 g/L; PLT  $\leq$  100 x 10<sup>9</sup> /L; HGB  $\leq$  110 g/L or PLT  $\leq$  100 x 10<sup>9</sup> /L; Any of above)

#### 10.5 **Treatment and Medications**

#### 10.5.1 **Prior Anticancer Therapies**

A prior anticancer therapy is defined as plasmapheresis or a systemic therapy subjects received, either as a single or combination therapy, for the treatment of WM with an end date occurring before the date of first dose of study treatment. Therapies given as a consolidation or maintenance of a response or remission will not be considered as a separate regimen. The number of lines and type of prior therapy for WM will be summarized.

#### 10.5.2 **Concomitant Medications**

Concomitant medications are defined as medications (any prescription or over-thecounter preparations, including vitamins and supplements) that were taken between 21 days before the date of the first dose of study drug and 30 days after the last dose of study drug. Concomitant medications after enrollment will be summarized by the World Health Organization (WHO) drug dictionary preferred term (PT).

#### 10.5.3 **Exposure to Study Drug**

Descriptive statistics (n, mean, standard deviation, median, and range) will be used to summarize:

- Duration of exposure (the interval between first dose date and last dose date)
- Actual cumulative dose administered (the total dose administered during the drug exposure period)
- Average daily dose (the ratio of actual cumulative dose administered and duration of exposure)
- Relative dose intensities (the ratio of actual cumulative dose to the planned cumulative dose)

A summary table that included number of subjects (and reasons) who had any dose withheld (any missed dose >= 7 days), and number of subjects (and reasons) who had

Acerta Pharma 

any dose reduction (any dose < 200 mg per day for >= 3 consecutive days) will be generated.

### 10.6 Analyses of Efficacy Endpoints

# 10.6.1 Definition of Primary Endpoints

ORR is defined as the proportion of subjects achieving a best overall response of either complete remission (CR), very good partial response (VGPR), partial response (PR), or MR before initiation of new anticancer therapy.

# 10.6.2 Analysis Method for Primary Endpoints

ORR will be estimated as the proportion of responders based on the best overall response. The 2-sided 95% CI will be calculated for ORR based on exact method. No formal statistical tests are performed for ORR.

Descriptive statistics will be provided for best overall response. The major response rate defined as the proportion of subjects who achieve PR or better (CR, VGPR, PR) will also be presented similarly as ORR. The ORR summaries will be generated separately for Owen 2013 criteria and modified 3<sup>rd</sup> IWWM workshop criteria.

# 10.6.3 Definition of Secondary Endpoints

### Duration of Response

DOR is defined as the interval from the first documentation of CR, VGPR, PR or MR to the earlier of the first documentation of definitive PD or death from any cause. DOR will be evaluated by IRC and investigator. Data from surviving, non-progressing subjects will be censored according to rules as documented in table 13.3.1 in appendix.

### Progression-free Survival

Progression-free survival (PFS) is defined as the interval from the start of acalabrutinib therapy to the earlier of the first documentation of definitive PD or death from any cause. Data from surviving, non-progressing subjects will be censored according to rules as documented in table 13.3.1 in appendix.

#### Overall Survival

The duration of overall survival (OS) will be measured from the start of acalabrutinib therapy until the date of death from any cause. Subjects who are known to be alive as

Acerta Pharma 

their last known status will be censored at their last date known to be alive. The censoring rule are documented in table 13.3.2 in appendix.

Patient Reported Outcome (PRO) --- EORTC QLQ-30

The EORTC QLQ-30 v3.0 will be used to assess the health-related quality of life. The EORTC QLQ-C30 v3.0 includes 30 separate items resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The scoring details are documented as:

| Domain | Scale | Number of<br>Items | Item<br>Range* | Component/Question<br>Item Numbers |
|---|---|---|---|---|
| Global health status/QoL | | | | |
| Global health status/QoL | QL2 | 2 | 6 | 29,30 |
| Functional scales | | | | |
| Physical functioning | PF2 | 5 | 3 | 1 to 5 |
| Role functioning | RF2 | 2 | 3 | 6, 7 |
| Emotional functioning | EF | 4 | 3 | 21 to 24 |
| Cognitive functioning | CF | 2 | 3 | 20, 25 |
| Social functioning | SF | 2 | 3 | 26, 27 |
| Symptom scales / items | | | | |
| Fatigue | FA | 3 | 3 | 10, 12, 18 |
| Nausea and vomiting | NV | 2 | 3 | 14, 15 |
| Pain | PA | 2 | 3 | 9,19 |
| Dyspnea | DY | 1 | 3 | 8 |
| Insomnia | SL | 1 | 3 | 11 |
| Appetite loss | AP | 1 | 3 | 13 |
| Constipation | СО | 1 | 3 | 16 |
| Diarrhea | DI | 1 | 3 | 17 |
| Financial difficulties | FI | 1 | 3 | 28 |

<sup>\*</sup> item range is the difference between the possible maximum and the minimum response to individual items;

From item 1 to 28 are scored as follows with the lower score indicates better quality of life: 1=not at all; 2=a little bit; 3=quite a bit; 4=very much. Item 29 and 30 are scored from 1 to 7, with 1 indicates very poor and 7 indicates excellent.

# 10.6.4 Analysis Method for Secondary Endpoints

ORR by IRC

Acerta Pharma 

Secondary analysis including the ORR evaluated by IRC based on modified 3rd IWWM workshop criteria. Summary table will be provided in the similar ways as specified in section 10.6.2.

### DOR

Kaplan-Meier method will be used for DOR analysis. KM estimates with 95% Cls will be calculated for event time quartiles, and event-free rates will be calculated at selected timepoints. The analysis will be generated separately for Owen 2013 criteria and modified 3<sup>rd</sup> IWWM workshop criteria. In addition, a listing for DOR will be generated including the reason for censoring. Only a subset of subjects will be included in DOR analysis.

#### PFS

The analysis of PFS is similar as DOR. A listing of PFS will be generated including the reason for censoring.

#### Overall Survival

The analysis of OS is similar as DOR. A listing of OS will be generated including the reason for censoring.

For all scales, the raw score (RS) is the mean of the component items:

raw score = RS = 
$$(I_1 + I_2 + \cdots + I_n)/n$$

For functional scales:

$$score = \left(1 - \frac{RS - 1}{range}\right) \times 100$$

For symptom scales/ items and global health status/QoL:

$$score = \left(\frac{RS - 1}{range}\right) \times 100$$

If at least half of the items from the scale been answered, use all the items that were completed and apply the standard equations above for calculating the scale scores. Ignore any items with missing values when making the calculation. If more than half of

Acerta Pharma 

the items from the scale is missing, the scale score is set as missing. For single-item measures, set score to missing if item is missing. The analysis windows for PRO scores are defined in table 10.4 at appendix.

At each assessment point, summary statistics of absolute and changes from baseline scale scores will be calculated. Summary tables of these statistics will be generated for all-treated population and a subset of subjects who achieve MR or better.

A listing of scale scores will be generated. A mean overtime plot will be generated for the global health status/quality of life.

#### 10.7 **Analyses Safety Endpoints**

#### 10.7.1 **Adverse Events**

The Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 will be used to code all AEs to a system organ class (SOC) and a PT. Subject incidence of the following events will be tabulated by SOC and PT in descending order of frequency through the AE reporting period. Summaries will also be presented by the severity of the AE (per common terminology criteria for adverse events [CTCAE], Version 4.03 or higher) and by relationship to study drug. Treatment emergent adverse event data will be summarized unless specified otherwise.

- treatment-emergent AEs
- treatment-emergent serious adverse events (TESAEs)
- treatment-related TEAEs
- treatment-related TESAEs
- AEs leading to study drug discontinuation or dose modifications or dose delay

Death summary table and a listing will be provided.

#### 10.7.2 **Adverse Events of Clinical Interest**

AEs of clinical interest are defined in section 8.5.1 of the SAP for acalabrutinib integrated summary of safety dated 21March2017.

Subject incidence rates of AEs of clinical interest will be tabulated using the CTCAE Version 4.03 or higher.

Acerta Pharma 

# 10.7.3 Laboratory Test Results

Laboratory data of hematology, serum chemistry, serum immunoglobulin, and T/B/NK cell count up to 30 days after last dose or the safety follow-up visit date, whichever is later, will be reported in SI units. Applicable laboratory results will be graded according to CTCAE Version 4.03 or higher. Generic normal ranges specified in American Medical Association (AMA) Manual of Style 10<sup>th</sup> Edition (2017) will be applied whenever reference ranges are not available.

Shift from baseline to worst grade during the treatment will be provided as shift tables for selected parameters. Figures of selected parameter will be plotted overtime as appropriate.

Figures of absolute values from baseline will be generated to assess effect of acalabrutinib on peripheral T/B/NK cell counts and on serum immunoglobulin levels.

### 10.7.4 Vital Signs

Summary statistics (mean, standard deviation, median, and range) will be produced for vital signs at baseline, maximum, change from baseline to maximum, last value, and change from baseline to last value.

To be included in the table, a subject must have both a baseline value and a postbaseline value for the given post-baseline time point.

### 10.7.5 Eastern Cooperative Oncology Group (ECOG) Performance Status

Change of ECOG from baseline to the maximum score up to 30 days after last dose or the safety follow-up visit date, whichever is later will be provided as shift tables.

# 10.7.6 Electrocardiogram (ECG)

ECG data is collected at screening. The investigator assessment of clinical significance categorized as normal, abnormal but not clinically significant, and abnormal clinically significant will be summarized. The number of subjects with corrected QT interval (QTc) greater than 480 msec will also be provided. A listing of subject with abnormal and clinically significant baseline ECG results or QTc> 480 msec will be produced.

#### 11. CHANGES FROM PROTOCOL-SPECIFIED ANALYSES

There is no major change from protocol-specified analyses.

Acerta Pharma 

# 12. LITERATURE CITATIONS / REFERENCES

Owen RG, Kyle RA, Stone MJ, et al. Response assessment in Waldenström macroglobulinaemia: update from the VIth International Workshop. BJH 2013;160:171-176.

Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, USDHHS, NIH, NCI; publish date May 28, 2009 (v4.03: June 14, 2010).

AMA Manual of Style 10th Edition. SI Conversion Calculator. Table 2. Selected Laboratory Tests, With Reference Ranges and Conversion Factors.

Steven P. Treon, Christina K. Tripsas, et al. Ibrutinib in Previously Treated Waldenström's Macroglobulinemia. N Engl J Med 2015 Oct 29;372(15):1430-1440.

EORTC QLQ-C30 Scoring Manual, 3<sup>rd</sup> Edition 2001, EORTC, Brussels. ISBN 2-9300 64-22-6.

Acerta Pharma 

### 13. APPENDICES

#### 13.1 Definitions

# **13.1.1** Study Day

The study day will be calculated refer to the date of first dose date. Study Day 1 is defined as the date of first dose of study drug. For assessments that occur on or after first dose date, study day is defined as (date of assessment – date of first dose + 1). For assessments that occur prior to first dose date, study day is defined as (date of assessment – date of first dose).

#### 13.1.2 Baseline Value and Post-baseline Value

Unless otherwise specified, the baseline value is defined as the last measurement taken on or prior to the first dose of study drug.

Change from baseline = Postbaseline value - Baseline value

Percentage change from baseline = 
$$\left(\frac{\text{change from baseline}}{\text{baseline}}\right) \times 100\%$$

# 13.1.3 Duration of Treatment and Time on Study

Duration of treatment will be calculated from the date of the first dose of study drug to the date of the last dose of study drug:

Duration of treatment = (last study drug date - first study drug date) + 1

Time on study will be calculated from the date of the first dose of study drug to the date of study exit or analysis data cut-off date, whichever is the earliest.

Time on study = (study exit date/data cut date - first study medication date) + 1

# 13.1.4 Average Daily Dose and Relative Dose Intensity

Average Daily Dose (mg/day) = Total cumulative dose taken (mg)/Duration of treatment

Relative Dose Intensity = 
$$\left(\frac{\text{Total cumulative dose taken}}{\text{Total expected dose}}\right) \times 100\%$$

where:

Total cumulative dose taken

= sum of actual daily dose taken through the duration of treatment;

Total expected dose = Duration of treatment  $\times$  Protocol assigned daily dose

Acerta Pharma 

# 13.1.5 Age

Age in years will be calculated at the date of enrollment.

#### 13.1.6 Year and Month

One year equals to 365.25 days and 1 month equals to 30.4375 days.

#### 13.1.7 Treatment-emergent Adverse Events

Treatment-emergent AEs are defined as those events that occur (actual or imputed start date) on or after the first dose of study drug, through the treatment phase, and within 30 days following the last dose of study drug.

# 13.1.8 Refractory Disease

Refractory disease will be categorized as "yes", "no" based on eCRF.

# 13.1.9 Extrameduallary Disease, Bone Marrow Involvement and Advanced Disease at Baseline

Data reported on 'bone marrow biopsy and aspirate' CRF will be used to derive bone marrow involvement. Subjects with bone marrow involved "positive" box checked at baseline will be considered to have bone marrow involved at baseline.

Data reported on 'tumor assessment prompt' CRF will be used to drive extrameduallary disease. Subjects with extrameduallary disease "yes" checked at baseline will be considered to have extrameduallary disease.

Subjects with either bone marrow involvement and/or extrameduallary disease at baseline will be considered to have advanced disease.

# 13.2 Imputation Rules for Partial or Missing Dates

Imputation of partial dates will be made for AE onset and stop dates, start and end dates of concomitant medication, start date of subsequent anticancer therapy, date of initial diagnosis and death date. If dates are completely missing, no imputation will be made. For any partial date with missing year, no imputation will be made.

The general rule for imputation is:

If only day is missing, then the 15<sup>th</sup> of the month will be used.

Acerta Pharma 

If only year is present, then June 30<sup>th</sup> will be used.

If such imputation date for initial diagnosis is on or after date of first dose, the date of first dose – 1 will be used. If such imputed date for subsequent anticancer therapies is before date of last dose, the date of last dose + 1 will be used.

If the imputed date is for an AE start date and is in the same year and month as the first dose date but before the first dose date, the first dose date will be used, or if the imputed AE start date is after the AE end date, the AE end date will be used. If the imputed date is for an AE start date and is in the same year and month as but after the last dose date + 30 days, the last dose date + 30 days will be used.

If the imputed date is for an AE end date and is after the death date, the death date will be used, or if the imputed AE end date is before the AE start date, the AE start date will be used.

For the missing death dates, if death year and month are available but day is missing:

- If mmyyyy for last contact date = mmyyyy for death date, set death date to the day after the last contact date.
- If mmyyyy for last contact date < mmyyyy for death date, set death date to the first day of the death month.
- If mmyyyy for last contact date > mmyyyy for death date, data error and do not impute.

If both month and day are missing for death date or a death date is entirely missing, do not impute and censor the subject survival time.

#### 13.3 **Censoring Rules**

The censoring rules for the DOR and PFS are documented in table 13.3.1.

Acerta Pharma 

Table 13.3.1 Censoring Rules for DOR and PFS

| Situation | Outcome | Event Description/ Censoring Reason | Last Analysis Date for DOR/PFS |
|---|---|---|---|
| Documented PD+ before initiation of new anticancer therapy or on/before data cutoff date, whichever occurred first | Event | PD | Earliest date of documented PD |
| Death without documented PD and not receiving new anticancer therapy on or before data cutoff | Event | Death | Date of Death |
| Documented PD or death after new anticancer therapy and the new anti-cancer started before data cutoff date | Censored | New anticancer<br>therapy | Date of last lack of PD* assessment on or prior to initiation of new anticancer therapy |
| No documented PD or death at the time of data cutoff and new anticancer therapy started before the data cutoff | Censored | New anticancer<br>therapy | Date of last lack of PD assessment on or prior to initiation of new anticancer therapy |
| Documented PD or death after new anticancer therapy and the new anticancer therapy started after data cutoff date | Censored | Data cutoff | Date of last lack of PD*<br>assessment on or before<br>data cutoff date |
| No documented PD or death<br>and subject not received new<br>anti-cancer therapy or new<br>anti-cancer therapy started<br>after the data cutoff | Censored | Data cutoff | Date of last lack of PD assessment on or before data cutoff |
| Withdrew consent without documented PD or death | Censored | Withdrew<br>consent | Date of last lack of PD assessment before withdrew or on/before data cutoff date whichever occurred first |

<sup>\*</sup> If multiple PD appears, the last lack of PD assessment refers to the last lack of earliest PD assessment.

The censoring rules for the OS are documented in table 13.3.2.

Table 13.3.2 Censoring Rules for OS

| Situation | Outcome | Event Description<br>or Censoring<br>Reason | Last Analysis Date for OS |
|---|---|---|---|
| Death on/before analysis data cutoff date | Event | Death | Death date |
| Patient alive on/before analysis data cutoff date | Censored | On-going | Date of last known alive |
| Not known to have died on/before analysis data cutoff date | Censored | Lost follow up | Date last known alive before analysis data cutoff date |
| Death after analysis data cutoff date | Censored | Death | Date of analysis data cutoff |

Acerta Pharma 

<sup>+</sup>All the PDs mentioned in SAP refer to confirmed PD as specified per protocol.

# 13.4 Analysis Windows for EORTC QLQ-30

The analysis windows for EORTC QLQ-30 is documented in table 13.4. In the case that more than 1 score is found with a time window, the score closest to the window center will be used in the analysis. In the case that there are 2 values that are equidistant from the center, the value prior to the center will be used.

**Table 13.4 Analysis Windows for EORTC QLQ-30** 

| Cycle | Study Day | Windows |
|-----------------|----------------|---------------------------------|
| Baseline | study day 1 | Day ≤ 1 |
| Cycle 2 Day 28 | study day 56 | 21 < Day ≤ 84 |
| Cycle 4 Day 28 | study day 112 | 84 < Day ≤ 140 |
| Cycle 6 Day 28 | study day 168 | 140 < Day ≤ 210 |
| Cycle 9 Day 28 | study day 252 | 210 < Day ≤ 294 |
| Cycle 12 Day 28 | study day 336 | 294 < Day ≤ 378 |
| Cycle 15 Day 28 | study day 420 | 378 < Day ≤ 462 |
| Cycle 18 Day 28 | study day 504 | 462 < Day ≤ 546 |
| Cycle 21 Day 28 | study day 588 | 546 < Day <= 630 |
| Cycle 24 Day 28 | study day 672 | 630 < Day <= 714 |
| Cycle 27 Day 28 | study day 756 | 714 < Day <= 798 |
| Cycle 30 Day 28 | study day 840 | 798 < Day <= 882 |
| Cycle 33 Day 28 | study day 924 | 882 < Day <= 966 |
| Cycle 36 Day 28 | study day 1008 | 966 <day <="1050&lt;/td"></day> |
| Cycle 39 Day 28 | study day 1092 | 1050 < Day <= 1134 |
| Cycle 42 Day 28 | study day 1176 | 1134 < Day <= 1218 |
| Cycle 45 Day 28 | study day 1260 | 1218 < Day <= 1302 |
| Cycle 48 Day 28 | study day 1344 | 1302 < Day <= 1386 |

Acerta Pharma 